CLINICAL TRIAL: NCT01594112
Title: Inappropriate Therapies and Home Monitoring® in Implantable Cardioverter Defibrillators (ICD)
Brief Title: Ability of Home Monitoring® to Detect and Manage the Inappropriate Diagnoses in Implantable Cardioverter Defibrillators.
Acronym: THORN
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: HS056
Record Dates: First submitted 2012-05-03; First posted 2012-05-08 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: ICD; Sudden Cardiac Death; Ventricular Fibrillation; Atrial Fibrillation; Ventricular Tachycardia
Keywords: Remote monitoring; Home monitoring; Defibrillators, Implantable cardioverter-defibrillator; Shock; Inappropriate diagnoses and Therapies; Corrective actions; ID recurrences; Medical reaction time
MeSH Terms: conditions — Death, Sudden, Cardiac; Ventricular Fibrillation; Atrial Fibrillation; Tachycardia, Ventricular; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with at least one ID: Patient with ICD who received at least one inappropriate diagnosis (with or without therapy) during the 15 months follow-up.

SUMMARY:
The purpose of the THORN registry is to show the ability of Home-Monitoring® to early identify and manage the inappropriate diagnoses of ventricular arrhythmia in ICD patients (i.e. lead rupture, atrial arrhythmia, oversensing…) whatever the type of device (single, dual, or triple chamber).

The electromyograms (iEGMs) provided by Remote Patient Monitoring will help the physician to early detect inadequate arrhythmia detection (ID) that can be responsible for inappropriate therapies (IT), and to take preventive actions in order to reduce the burden of these inappropriate therapies.

THORN is an observational epidemiologic, prospective and multicenter registry. The primary objective is to measure the relative proportion of patients experiencing at least one inappropriate therapy during a fifteen months follow-up period. Moreover, THORN will assess the incidence, predictors, outcome and recurrence of inappropriate diagnoses in 1750 ICD patients.

DETAILED DESCRIPTION:
Remote Patient Monitoring allows early detection of events that can generate inadequate detection of ventricular arrhythmia (i.e. lead rupture, atrial arrhythmia, oversensing….) and be responsible for inappropriate therapies. In such cases, it may be assumed that physicians can react earlier and take preventive actions, in order to reduce the risk or burden of inappropriate therapies.

The THORN registry has two purposes:

* To determine retrospectively the relative proportion of patients experiencing at least one inappropriate therapy during 15-months of follow-up, in ICD patients equipped with Home Monitoring®. This part concern 1240 patients.
* To evaluate prospectively the relationship between the detection of inappropriate diagnosis (with or without subsequent inappropriate therapy), the corrective action taken, and the recurrences of inappropriate diagnosis of the same origin/mechanism. This part concerns 510 patients.

BIOTRONIK Home Monitoring® by iEGM-Online® with Biotronik ICD devices (LUMAX) systematically stores any episode classified as ventricular tachycardia (VT) or ventricular fibrillation (VF) which is transmitted to the physician.

In the THORN study, in addition to the physicians' analysis, all electromyograms will be reviewed by an adjudication committee in order to classify them as appropriate or inappropriate diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject implanted with a single, dual, or triple chambers ICD within the last 3 months
* Home Monitoring® activated and functional since hospital discharge
* Patient willing and able to comply with the protocol and who has provided written informed consent about Home Monitoring®,
* Patient whose medical situation is stable

Exclusion Criteria:

* ICD replacements
* New York Heart Association Function Class IV patients
* Pregnant women or women who plan to become pregnant during the trial
* Presence of any disease, other than patient's cardiac disease, associated with reduced likelihood of survival for the duration of the trial, e.g. cancer, uraemia (urea > 70mg/dl or creatinine >3mg/dl), liver failure, etc.
* Age < 18 years
* Patient unable to handle the Biotronik's transmitter correctly
* Change of residence expected during the study
* Insufficient global system for mobile communication (GSM) coverage at patient's home
* Participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population implanted of ICD with Biotronik Home Monitoring® system. 512 patients will be selected by investigators in 50 centers in France.
Sampling Method: Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2012-03-15 (Actual); Primary Completion 2013-09-27 (Actual); Study Completion 2015-04-01 (Actual)

PRIMARY OUTCOMES:
Relative proportion of patients experiencing at least one inappropriate therapy (retrospective part) or more than one inappropriate therapy (prospective part) | 15 months
  Study of the relationship between the detection of ID, the corrective action taken and the recurrence of ID of the same mechanism.

SECONDARY OUTCOMES:
Number of diagnoses per patient per year and relative proportion of patients with at least one diagnosis | 15 months
  The number of diagnoses per patient per year and the associated proportion of patients (with at least one diagnosis) will be measured. This will give the incidence rate of experiencing special classes of diagnoses over the 15-months follow-up period. The following subclasses will be assessed:
  Appropriate or not diagnoses, ID without therapy, therapies defined as shocks or antitachycardia pacing (ATP), shocks, inappropriate shocks, recurrence of ID and recurrence of inappropriate shocks.
  The prospective part will be compared to the retrospective part.
Relative proportion of patients with a second day of ID | 15 months
  Knowing that the intervals between ID days cannot be predetermined (non normal distribution), medical reaction time anticipated with Home Monitoring® can reduce the number of patients with a second day of ID.
  The proportion of patients with more than one inappropriate diagnosis will be measured.
Number of Asymptomatic Inappropriate therapy and Inappropriate therapy without diagnosis | 15 months
  Knowing that the main added value of Home Monitoring® relates on asymptomatic inappropriate therapies and inappropriate diagnoses without therapy (IDWT), the number of asymptomatic IT or IDWT patient per year and the associated proportion of patients (with at least one inappropriate diagnosis) will be measured.
Time to the first ID | 15 months
  The time from the enrolment until the first EGM revealing the ID will be assessed.
Medical reaction time to the ID | 15 months
  The time from the first ID to the follow-up visit during which a corrective action is taken is defined as the medical reaction time and will be assessed.
  In case of hospitalization without a follow-up visit (lead replacement for instance), the first day of hospitalization will be considered as the follow-up visit date.
  In current practice, the patients receiving shocks are advised to call their physicians in order to have their ICD interrogated. The analysis will distinguish the symptomatic IT and the asymptomatic ID (asymptomatic IT or IDWT).
Number of days of recurrence within the medical reaction time | 15 months
  The number of days with at least one ID within the medical reaction time is defined as the number of days of recurrence and will be evaluated with the associated proportion of patients. The analysis will distinguish the symptomatic IT and the asymptomatic ID (asymptomatic IT or IDWT).
Effectiveness of the corrective action and analysis according to the initial ID type | 15 months
  The proportion of patients with at least one inappropriate diagnosis recurrence (first day of recurrence) after the corrective action, and with the same ID mechanism as the original one, will be evaluated.
  A subgroup analysis depending on the ID mechanism will be performed, considering the inhomogeneous efficiency of the corrective action depending on the initial mechanism of the inappropriate diagnosis/therapy .
  The time from the follow-up visit during which the corrective action is taken until the next ID will be measured to assess the effectiveness of the corrective action.
Classification of ID | 15 months
  The proportion of patient in the following classes of ID episodes will be evaluated:
  * Atrial fibrillation,
  * Other forms of supraventricular tachyarrhythmia
  * Sinus tachycardia
  * Abnormal sensing (T wave oversensing, interferences,…)
  * Other: the comparison is performed as an inter observer comparison between the Adjudication Board's and the physician's classification.
Total number of hospitalizations/deaths related to ID and IT | 15 months
  Knowing that inappropriate therapies are among the heaviest ICD side-effects, the total number of hospitalizations and deaths related to ID or IT will be assessed.
Risk of all-cause mortality | 15 months
  The risk of death associated with inappropriate therapy only, with the inappropriate shocks only, with any shocks, without any therapy, without any shocks will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude DEHARO, Pr. Dr., Principal Investigator — Hôpital La Timone, 264 rue St. Pierre, 13385 MARSEILLE Cedex 5
Locations (55):
- France (55):
  - CH d'Aix en Provence, Aix-en-Provence
  - CH d'Angers, Angers
  - CH d'Avignon, Avignon
  - CH de la Cote Basque, Bayonne
  - Clinique Lafourcade, Bayonne
  - Clinique Saint Augustin, Bordeaux
  - CHU de Nancy, Bourgogne
  - CHU la Cavale Blanche, Brest
  - CH William-Morey, Chalon-sur-Saône
  - CHG de Chateauroux, Châteauroux
  - Hôpital Militaire, Clamart
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Albert Schweitzer, Colmar
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CH de DAX, Dax
  - CHU de Dijon, Dijon
  - CHU Albert Michalon, Grenoble
  - CH de Haguenau, Haguenau
  - CH de Lagny sur Marne, Lagny-sur-Marne
  - CH Robert Boulin, Libourne
  - CHRU de Lille, Lille
  - CH St Luc St Joseph, Lyon
  - Clinique de la Sauvegarde, Lyon
  - Hôpital Cardiologique, Lyon
  - Hôpital Nord, Marseille
  - Hôpital La Timone, Marseille
  - Institut Jacques Cartier, Massy
  - CHI de Montfermeil, Montfermeil
  - CHU de Montpellier, Montpellier
  - Clinique du Milénaire, Montpellier
  - CH de Moulins, Moulins
  - Clinique Ambroise Paré, Nancy
  - CHU G. & R. Laënnec, Nantes
  - CHU Nîmes, Nîmes
  - Hôpital Georges Pompidou, Paris
  - CH de Pau, Pau
  - Clinique Saint Pierre, Perpignan
  - CHU Bordeaux, Pessac
  - CH de Périgueux, Périgueux
  - CHU la Mileterie, Poitiers
  - CHU (Hôpital Pontchaillou), Rennes
  - CH de Rodez, Rodez
  - Chu Hôpital Charles Nicolle, Rouen
  - CH de Saint Brieuc, Saint-Brieuc
  - CHU de St-Etienne, Saint-Etienne
  - CH d'Angoulême, Saint-Michel
  - Hôpital Font Pré, Toulon
  - Clinique Pasteur, Toulouse
  - CHRU Tours (Hôpital Trousseau), Tours
  - Clinique Saint Joseph, Trélazé
  - CH de Troyes, Troyes
  - CH de Valence, Valence
  - CH de Valenciennes, Valenciennes
  - CH Bretagne Atlantique, Vannes
  - CH de Villefranche, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perrin T, Boveda S, Defaye P, Rosier A, Sadoul N, Bordachar P, Klug D, Ritter P, Belhameche M, Babuty D, Mansourati J, Lazarus A, Deharo JC. Role of medical reaction in management of inappropriate ventricular arrhythmia diagnosis: the inappropriate Therapy and HOme monitoRiNg (THORN) registry. Europace. 2019 Apr 1;21(4):607-615. doi: 10.1093/europace/euy284. PMID 30605510